CLINICAL TRIAL: NCT06343337
Title: The Effects of Pregnancy on Oral Health, Salivary ph and Flow Rate
Brief Title: The Effects of Pregnancy on Oral Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Fatma Yilmaz, Asistant Professor, Muğla Sıtkı Koçman University
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: MSKUDİSCLİNİCALTRİALS_FYİLMAZ.
Record Dates: First submitted 2024-02-29; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Pregnancy Related; Dental Caries; Periodontal Diseases; Saliva Altered
Keywords: CPI; DMFT; Unsitumulated saliva; Pregnant woman
MeSH Terms: conditions — Dental Caries; Periodontal Diseases | interventions — Gravidity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The individual who evaluates the salivary pH and flow rate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- First trimester (Experimental)
  Interventions: Diagnostic Test: Evaluation of DMFT index, CPI scores, salivary pH and flow rate in pregnant and non-pregnant woman
- Second trimester (Experimental)
  Interventions: Diagnostic Test: Evaluation of DMFT index, CPI scores, salivary pH and flow rate in pregnant and non-pregnant woman
- Third Trimester (Experimental)
  Interventions: Diagnostic Test: Evaluation of DMFT index, CPI scores, salivary pH and flow rate in pregnant and non-pregnant woman
- Non-pregnant woman (Other): Control group
  Interventions: Diagnostic Test: Evaluation of DMFT index, CPI scores, salivary pH and flow rate in pregnant and non-pregnant woman

INTERVENTIONS:
Diagnostic Test: Evaluation of DMFT index, CPI scores, salivary pH and flow rate in pregnant and non-pregnant woman — Total 198 volunteer (51 women for control, 47 women for 1st trimester, 51 women for 2nd trimester, and 49 women for 3rd trimester) were included. The data about sociodemographic characteristics, dental and systemic health conditions were recorded. Unsitumulated saliva samples were collected for 5 minutes by spitting method. The pH of saliva was measured by a portable pHmeter. The salivary flow rate was determined by the weight measurement method. DMFT index and CPI scores were determined. The statistical differences were evaluated by Kruskal-Wallis, Mann Whitney U and Chi Square tests (α=.05).

SUMMARY:
The aim of this study was to evaluate the effects of pregnancy on salivary pH, flow rate, caries experience and periodontal status.

The main questions it aims to answer are:

* Does pregnancy affect caries experience and periodontal status?
* Does pregnancy affect salivary pH and flow rate?
* Is there a difference between pregnant and non-pregnant woman with respect to caries experience, periodontal status, salivary pH and flow rate?
* Is there a difference among first, second and third trimester with respect to caries experience, periodontal status, salivary pH and flow rate?

DETAILED DESCRIPTION:
The basic physiological changes that occur during pregnancy affect the oral health of women as well as their general health. Although it is thought that physiological and hormonal changes increase susceptibility to periodontal diseases and dental caries that are among the most common health problems in society, the results obtained from studies on this subject are controversial. The fact that women often encounter these diseases during pregnancy may be due to many factors such as accumulation of dental plaque, differentiation in microbial composition, changes in the amount of saliva, and decreases in pH.Increases in levels of steroid hormones, especially during pregnancy, decrease the resistance of the gingiva against periodontal pathogens, and increase gingival vascularity and blood flow, causing pregnancy gingivitis.

Dental caries is a multifactorial infectious disease characterized by mineral loss in dental hard tissues. In pregnancy, calcium loss occurs in the hard tissues of the teeth, similar to the bones, through the pulpal route, and the concentration of calcium and phosphate in the saliva also decreases. This increases demineralization in dental tissues and decreases remineralization.

Many environmental factors, such as nutrition, oral hygiene habits, socio-economic status, educational status, and the amount and quality of saliva, play some roles in the development of caries. It is thought that one reason dental caries is more common during pregnancy is changes in the amount and content of saliva. Although some studies have found that the salivary glands are affected by pregnancy, as in other exocrine glands, others have reported that the amount of saliva and its flow rate do not change significantly during this period.

In the literature, there are many controversial results regarding whether the amount and quality of saliva change with pregnancy, how they change in different trimesters of pregnancy, and how these changes affect tooth and periodontal diseases. For this reason, this study aimed to evaluate the salivary pH, flow rate, caries prevalence, and periodontal status of women in different trimesters of pregnancy and non-pregnant women.

2. Materials & Methods The experimental design was in accordance with the Consolidated Standards of Reporting Trials (CONSORT) statement.

2.1. Ethical Statement This study was conducted in accordance with the Principles of the Declaration of Helsinki. Ethical approval was received for this research from the Ethics Committee of Health Sciences of …………. University (Report no: 21/VII).

2.2. Participants Volunteer pregnant in different trimesters (for study groups) and non-pregnant women (for control group) (18-35 ages) who applied to the Obstetrics and Gynecology Outpatient Clinic of the Faculty of Medicine of Mugla Sitki Kocman University were included in this study. Their written informed consent was obtained before they took part. Individuals with severe systemic disease, those who used drugs that directly affect salivary flow rate (e.g., antihypertensive, diuretic, psychotherapeutic, and antiarthritic medications), and those who used cigarettes or alcohol were excluded from the study.

2.3. Study size The G*Power package program was used to perform a power analysis to determine the sample size. At 95% confidence level 80% power was obtained with at least 128 samples for f=0.3 effect size (n=32). In this context, we aimed to reach minimum 45 participants for each group.

2.4. Data sources/ measurement Questions were asked about participants' sociodemographic characteristics, systemic health conditions, eating habits, dental care routines, and oral and dental problems, and the data were recorded. To evaluate the salivary flow rate and pH, the unstimulated saliva of the participants was collected at least 1 hour after breakfast, between 10:00 and 11:00 in the morning, at 23°C room temperature with 61.5% humidity for 5 minutes, using the spitting method. Before beginning the saliva collection process, those who felt hungry or thirsty were allowed to drink water and eat, but then participants were asked to brush their teeth, and saliva collection was started 1 hour later. During sample collection, individuals were allowed to sit in a comfortable position, with their head forward and mouth slightly open, and they were asked not to speak. Samples were collected in sterile, dry, pre-weighted deionized glass test tubes. The pH analysis was performed using a calibrated benchtop pH meter (Hanna Instruments®, HI 2211, Woonsocket, RI, USA) within half an hour of sample collection to prevent degradation of the saliva. The salivary flow rate was determined by the weight measurement method using sensitive scales (Shimadzu, AW220, Japan). To determine the net saliva amount, the tare weight of the container tube was subtracted from the saliva-filled gross weight and divided by 5, and the flow rate per minute was determined in g/min or l/min considering the salivary density equal to 1 g/cm3 with an uncertainty of ± 0.001 rpm. (Flow Rate = Gross Weight-Tare Weight/5 min). The obtained data were recorded.

The caries experience and periodontal status of the participants were determined by a dentist who had undergone standardization and calibration training in accordance with the recommendations and criteria of the World Health Organization. Caries experience was measured by the DMFT index (total number of decayed, missing, and filled teeth). The Community Periodontal Index (CPI) values used to determine periodontal health status were scored between 0 and 4 (0: health periodontal conditions; 1: gingival bleeding on probing; 2: calculus and bleeding; 3: periodontal pocket 4-5 mm; and 4: periodontal pocket ≥5.5 mm ) were determined.

2.5. Statistical methods For statistical evaluation, SPSS software version 25.0 (IBM, Armonk, NY: IBM Corp.) was used. Data were first evaluated using the Kolmogorov-Smirnov and Shapiro-Wilk tests to evaluate distribution normality. Thereafter, the Kruskal-Wallis test (post hoc: Mann-Whitney U test with Bonferroni correction) and Mann-Whitney U test were used to test the statistical differences among groups for continuous variables. Chi square and Fisher exact tests were used to test the statistical differences among groups for categorical variables. Spearman's correlation coefficient was used to examine the correlation between continuous variables (α=.05).

ELIGIBILITY:
Inclusion Criteria for study arms

* Volunteer participants
* Pregnant women aged 18-35 years
* Pregnant woman in different trimesters
* Those who applied to Muğla Sıtkı Koçman University Faculty of Medicine Gynecology and Obstetrics Outpatient Clinic

Inclusion Criteria for control arm

* Volunteer participants
* Non-pregnant women aged 18-35 years
* Those who applied to Muğla Sıtkı Koçman University Faculty of Medicine Gynecology and Obstetrics Outpatient Clinic

Exclusion Criteria:

* Individuals with severe systemic disease
* Individuals who used drugs that directly affect salivary flow rate (e.g., antihypertensive, diuretic, psychotherapeutic, and antiarthritic medications)
* Individuals who used cigarettes or alcohol

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant and non-pregnant woman
Enrollment: 198 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
The effects of pregnancy on caries experience | Five minutes after the saliva sample was collected.
  DMFT index was determined according to the sum of the number of decayed, missing and filled teeth according to WHO criteria.
The effects of pregnancy on periodontal status. | Five minutes after the saliva sample was collected.
  The Community Periodontal Index (CPI) values used to determine periodontal health status were scored between 0 and 4 (0: health periodontal conditions; 1: gingival bleeding on probing; 2: calculus and bleeding; 3: periodontal pocket 4-5 mm; and 4: periodontal pocket ≥5.5 mm ) were determined.
The effects of pregnancy on salivary pH. | Salivary pH measurements were made within half an hour at the latest after the saliva samples were taken.
  To evaluate the salivary pH, the unstimulated saliva of the participants was collected. The pH analysis was performed using a calibrated benchtop pH meter (Hanna Instruments®, HI 2211, Woonsocket, RI, USA) within half an hour of sample collection to prevent degradation of the saliva.
The effects of pregnancy on salivary flow rate. | Saliva flow rate measurements were made within half an hour at the latest after the saliva samples were taken.
  The salivary flow rate was determined by the weight measurement method using sensitive scales (Shimadzu, AW220, Japan). To determine the net saliva amount, the tare weight of the container tube was subtracted from the saliva-filled gross weight and divided by 5, and the flow rate per minute was determined in g/min or l/min considering the salivary density equal to 1 g/cm3 with an uncertainty of ± 0.001 rpm. (Flow Rate = Gross Weight-Tare Weight/5 min).

CONTACTS AND LOCATIONS:
Overall Officials: FATMA YILMAZ, Asistant Professor, Study Chair — Muğla Sıtkı Koçman Universty; Ozgul Carti Dorterler, Asistant Professor, Principal Investigator — Muğla Sıtkı Koçman Universty; Saniye Eren Halici, Asistant Professor, Principal Investigator — Muğla Sıtkı Koçman Universty; Burcu Kasap, Professor, Principal Investigator — Muğla Sıtkı Koçman Universty; Aysegul Demirbas, Professor, Study Director — Ege Universty
Locations (1):
- Fatma Yilmaz, Menteşe, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] Kateeb E, Momany E. Dental caries experience and associated risk indicators among Palestinian pregnant women in the Jerusalem area: a cross-sectional study. BMC Oral Health. 2018 Oct 22;18(1):170. doi: 10.1186/s12903-018-0628-x. PMID 30348139
- [Background] Kamate WI, Vibhute NA, Baad RK. Estimation of DMFT, Salivary Streptococcus Mutans Count, Flow Rate, Ph, and Salivary Total Calcium Content in Pregnant and Non-Pregnant Women: A Prospective Study. J Clin Diagn Res. 2017 Apr;11(4):ZC147-ZC151. doi: 10.7860/JCDR/2017/24965.9516. Epub 2017 Apr 1. PMID 28571283
- [Background] Srinivas SK, Parry S. Periodontal disease and pregnancy outcomes: time to move on? J Womens Health (Larchmt). 2012 Feb;21(2):121-5. doi: 10.1089/jwh.2011.3023. Epub 2011 Oct 12. PMID 21992584
- [Background] Wu M, Chen SW, Jiang SY. Relationship between gingival inflammation and pregnancy. Mediators Inflamm. 2015;2015:623427. doi: 10.1155/2015/623427. Epub 2015 Mar 22. PMID 25873767
- [Background] Laine MA. Effect of pregnancy on periodontal and dental health. Acta Odontol Scand. 2002 Oct;60(5):257-64. doi: 10.1080/00016350260248210. PMID 12418714
- [Background] Selwitz RH, Ismail AI, Pitts NB. Dental caries. Lancet. 2007 Jan 6;369(9555):51-9. doi: 10.1016/S0140-6736(07)60031-2. PMID 17208642
- [Background] Laine M, Tenovuo J, Lehtonen OP, Ojanotko-Harri A, Vilja P, Tuohimaa P. Pregnancy-related changes in human whole saliva. Arch Oral Biol. 1988;33(12):913-7. doi: 10.1016/0003-9969(88)90022-2. PMID 3256298
- [Background] Laine M, Pienihakkinen K. Salivary buffer effect in relation to late pregnancy and postpartum. Acta Odontol Scand. 2000 Feb;58(1):8-10. doi: 10.1080/000163500429361. PMID 10809393
- [Derived] Yilmaz F, Carti Dorterler O, Eren Halici S, Kasap B, Demirbas A. The effects of pregnancy on oral health, salivary ph and flow rate. BMC Oral Health. 2024 Oct 25;24(1):1286. doi: 10.1186/s12903-024-05057-0. PMID 39455976